CLINICAL TRIAL: NCT06434636
Title: The Effect of The Use of Low Dose Tranexamic Acid on Surgeon Satisfaction, Side Effects and Complications in Endoscopic and Microscopic Ear Surgery Cases Which Are Used With Controlled Hypotension
Brief Title: The Effect of Tranexamic Acid in Endoscopic and Microscopic Ear Surgery Cases on Surgeon Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Talha Ersoy, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024/88
Record Dates: First submitted 2024-05-19; First posted 2024-05-30 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Middle Ear Disease
Keywords: tranexamic acid; controlled hypotension; middle ear surgery
MeSH Terms: interventions — Tranylcypromine; Injections; Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups: Intervention (M) and Control (C). Just before the operation begins, 10 mg/kg tranexamic acid (TXA) will be administered to the intervention group in 100 mL of 0.9% physiological saline (SF) solution in 15 minutes. 100 mL of 0.9% SF solution will be sent to the control group in 15 minutes.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (I) (Active Comparator): Patients' vital values will be recorded before surgery.10 mg/kg tranexamic acid (Transamine 10% IV/IM Solution for Injection) is added into 100 cc serum through the appropriate vascular access and injected for 15 minutes.The amount of bleeding in the surgical field will be evaluated by the surgeon using the Boezaart Scale.Intraoperatively, hemodynamic changes such as bradycardia, tachycardia, arrhythmia and agents used such as vasopressors, antiarrhythmics and vagolytics will be recorded in the patient.Post-Operatively the surgeon's quality of vision will be questioned with the Surgeon Satisfaction Scale.Postoperative 0th, 12th, and 24th developments - the presence of vomiting and postoperative complaints will be questioned.The presence of bleeding or complications in the first 2 weeks after surgery will be questioned.The presence of thromboembolic events and other services will be questioned within 12 weeks after surgery.
  Interventions: Drug: Transamine 10% IV/IM Solution for Injection
- Control Group (C) (Placebo Comparator): Preoperative vital values of the patients will be recorded.100 cc of physiological saline will be sent through the appropriate vascular access in 15 minutes.
  The amount of bleeding in the surgical field will be evaluated by the surgeon using the Boezaart Scale. Intraoperatively, hemodynamic changes such as bradycardia, tachycardia, arrhythmia that develop in the patient, and agents such as vasopressors, antiarrhythmics, and vagolytics used will be recorded.
  Postoperatively the surgeon's quality of vision will be questioned with the Surgeon Satisfaction Scale. The presence of nausea and vomiting and postoperative complaints will be questioned at the 0th, 12th, and 24th postoperative hours. The presence of surgical bleeding or complications that occur in the first 2 weeks of surgery will be questioned. The presence of thromboembolic events and other complications will be questioned within 12 weeks postoperatively.
  Interventions: Drug: %0.9 Saline

INTERVENTIONS:
Drug: Transamine 10% IV/IM Solution for Injection — 10 mg/kg tranexamic acid (Transamine 10% IV/IM Injectable Solution) will be placed into 100 cc physiological saline through the appropriate vascular access and injected within 15 minutes.
  Other Names: tranexamic acid
  Arms: Intervention Group (I)
Drug: %0.9 Saline — 100 cc %0.9 Normal Saline will be injected through the appropriate vascular access within 15 minutes
  Other Names: Physiological Saline; %0.9 NaCl
  Arms: Control Group (C)

SUMMARY:
By using tranexamic acid, an antifibrinolytic drug, the aim is to prevent the restriction of the field of view of the surgical field due to bleeding in middle ear microscopic and endoscopic surgery operations in which controlled hypotension is applied, and therefore the prolongation of the surgical time, and to increase surgeon satisfaction.

DETAILED DESCRIPTION:
After obtaining approval from our university and the Turkish Ministry of Health's pharmaceutical and medical device agency and written consent from the patients, 100 patients who underwent middle ear surgery using controlled hypotension under general anesthesia will be included in the study.

The study will be conducted in a randomized controlled, double-blind manner. Patients between the ages of 18-65 and with American Society of Anesthesiologists (ASA) Scores I and II will be included in the study. Patients will be divided into two groups: Intervention (M) and Control (C). Just before the operation begins, 10 mg/kg tranexamic acid (TXA) will be administered to the intervention group in 100 mL of 0.9% physiological saline (SF) solution in 15 minutes. 100 mL of 0.9% SF solution will be sent to the control group in 15 minutes. At the end of the operation, the operator's quality of vision of the surgical field will be recorded by questioning the surgeon's satisfaction with the Boezaart Score and the Surgeon Satisfaction Score.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-65
* Individuals with ASA I (no additional disease) or ASA II (mild systemic disease)
* Those who do not have a disease such as thrombophilia or bleeding diathesis will be included in the study

Exclusion Criteria:

* Patients with ASA III (those with uncontrolled chronic disease) or above
* Patients with cardiovascular disease, congestive heart failure, coronary artery disease, cerebrovascular insufficiency, renal or hepatic failure
* Patients with thrombophilia, bleeding diathesis, coagulation defects
* Pregnant patients
* Those with a history of any allergic reaction to tranexamic acid and its derivatives will be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders will be included this study
Enrollment: 100 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
Boezaart et al grading scale | 2-3 hours
  At the end of a surgery, the surgical field was graded in terms of bleeding by the surgeon using the scale used by Boezaart et al in 1995;
  0 : No bleeding (cadaveric conditions).
  1. : Slight bleeding: no suctioning required.
  2. : Slight bleeding: occasional suctioning required.
  3. : Slight bleeding: frequent suctioning required. Bleeding threatens surgical field a few seconds after suction is removed.
  4. : Moderate bleeding: frequent suctioning required and bleeding threatens surgical field directly after suction is removed.
  5. : Severe bleeding: constant suctioning required; bleeding appears faster than can be removed by suction; surgical field severely threatened and surgery usually not possible.
Surgeon Satisfaction Score | 2-3 hours
  At the and of surgery , surgeon's satisfaction with surgical field quality was also graded in a 5-item Likert scale, where 1 = poor and 5 = excellent

CONTACTS AND LOCATIONS:
Overall Officials: Talha ERSOY, MD, Study Chair — TC Erciyes University
Locations (1):
- Erciyes Üniversitesi, Kayseri, Talas, Turkey (Türkiye)